CLINICAL TRIAL: NCT05640622
Title: Reliability and Validity of the Turkish Version of the Gait Outcomes Assessment List (GOAL) for Children With Cerebral Palsy
Brief Title: Turkish Validity and Reliability of Gait Outcomes Assessment List (GOAL)
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Umut Apaydin, PhD, PT, Principal Investigator, Gazi University
Other Study IDs: E-77082166-604.01.02-487509
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gait Outcomes Assessment List (GOAL) — Gait Outcomes Assessment List (GOAL) is a scale developed to contribute to the determination of treatment goals. This questionnaire includes the priorities, expectations, and goals of children with CP who can walk and reveals their walking characteristics.

SUMMARY:
The aim of this study is to investigate the reliability and validity of the Turkish Gait Outcomes Assessment List (GOAL) Questionnaire, in children with cerebral palsy (CP) with GMFCS level1, 2, and 3.

DETAILED DESCRIPTION:
Most children with cerebral palsy (CP) can walk. Musculoskeletal disorders of these children cause deterioration in gait functions. Disruptions in gait limit children's participation. To minimize these impairments, various interventions are usually applied to children with CP who can walk. The ultimate goal of these interventions is to help these children achieve the best possible participation in activities of daily living. In addition, goal determination by children and families in treatment planning is important in terms of treatment success. The Gait Outcomes Assessment List (GOAL) is a scale developed to contribute to the determination of these goals. This questionnaire includes the priorities, expectations, and goals of children with CP who can walk and reveals their walking characteristics. The questionnaire is used in two languages, English and German, and there is no Turkish version of the questionnaire. Therefore, the aim of this study is to create the Turkish version of the 'Gait Outcomes Assessment List (GOAL)' family and child questionnaires and to examine its validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy
* Being able to read and write Turkish

Exclusion Criteria:

* Children who have had botox or orthopedic surgery in the last 6 months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Cerebral Palsy with GMFCS level 1,2, and 3
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Gait Outcomes Assessment List (GOAL) | 2 weeks
  The GOAL consists of 49 items grouped into seven domains: domain A, activities of daily living and independence; domain B, gait function and mobility; domain C, pain, discomfort, and fatigue; domain D, physical activities, sports, and recreation; domain E, gait pattern and appearance; domain F, use of braces and mobility aids; and domain G, body image and self-esteem. Domains A, B, D, and E consist of 6-point Likert scales changing from extremely difficult to no problem at all. Domain C consists of 5-point Likert scales changing from everyday to none of the time. Domains F and G, consist of 5-point Likert scales changing from very unhappy to very happy. Domain and total GOAL scores were calculated for each child and ranged from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Functional Mobility Scale (FMS) | 2 weeks
  The FMS is a performance measure, classifying mobility on the basis of the use of mobility devices across three distances, 5m, 50m, and 500m, which represent home, school, and community distances. Assessment is by the clinician on the basis of questions asked of the parent or child. The mobility of the child is scored from 1 to 6 for each distance, with 1 representing the use of a wheelchair and 6 representing independence on all surfaces.
Gillette Functional Assessment Questionnaire (FAQ) | 2 weeks
  The Gillette Functional Assessment Questionnaire (FAQ) is a self or proxy-report measure that includes a ten-level classification of ambulatory function (FAQ Walking Scale), and 22 functional locomotor activities rated on a five-level Likert difficulty scale (FAQ 22-item skill set). The FAQ 22-item skill set includes common functional mobility activities that further characterize the individual's locomotor abilities. The five-level Likert response scale used for the 22 skill items was 'easy', 'a little hard', 'very hard', 'can't do at all', and 'too young for activity'.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thomason P, Tan A, Donnan A, Rodda J, Graham HK, Narayanan U. The Gait Outcomes Assessment List (GOAL): validation of a new assessment of gait function for children with cerebral palsy. Dev Med Child Neurol. 2018 Jun;60(6):618-623. doi: 10.1111/dmcn.13722. Epub 2018 Mar 24. PMID 29573409
- [Result] Bonfert MV, Jelesch E, Hartmann J, Koenig H, Warken B, Meuche A, Jung NH, Bernius P, Weinberger R, Sorg AL, von Kries R, Narayanan UG, Hoesl M, Berweck S, Schroeder AS. Test-Retest Reliability and Construct Validity of the German Translation of the Gait Outcome Assessment List (GOAL) Questionnaire for Children with Ambulatory Cerebral Palsy. Neuropediatrics. 2022 Apr;53(2):96-101. doi: 10.1055/s-0040-1722688. Epub 2021 Dec 21. PMID 34933378